CLINICAL TRIAL: NCT05220111
Title: Quality of Life 12 Months After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R12265
Record Dates: First submitted 2022-01-14; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Quality of Life
Keywords: Quality of Life, postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgical operation (valve, aorta, coronary arteries) — Quality of life assessment using EQ-5D-3L
  Other Names: Quality of life assessment

SUMMARY:
Cardiac surgical patients entering the hospital for operation were voluntarily recruited to participate a 12 month follow- up of health related quality of life (QOL)

DETAILED DESCRIPTION:
Cardiac surgical patients entering the hospital for operation were voluntarily recruited to participate a 12 month follow- up of health related quality of life based on established QOL measurements with EuroQol quality of life 5 dimensional 3 level (EQ-5D-3L) description system at preoperative, 6 months and 12 months postoperatively. The study started on May 2013 and ended at the end of 2018. The data has been analyzed for publication in 2021. The total number of patients reached 1594.

ELIGIBILITY:
Inclusion Criteria:

* elective or urgent cardiac surgery (open heart procedure to valves or ascending aorta /arch, on-pump or off-pump surgery to the coronary arteries )
* willingness to participate,
* ability to comprehend Finnish language

Exclusion Criteria:

* emergency surgery (with no time to introduce the study in good time)
* not willing to participate,
* blind or other disturbance in seeing,
* inability to comprehend Finnish language

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers for primary or secondary major cardiac surgery (cabg, valve, aorta or combined procedures)
Sampling Method: Non-Probability Sample
Enrollment: 1594 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
EQ-Visual Analogue Scale result, preoperative | preoperative
  EQ-Visual Analogue Scale, scale 0 (worst) to 100 (best possible), in percent
EQ-Visual Analogue Scale result, at 6 months | 6 months after surgery
  EQ-Visual Analogue Scale, scale 0 (worst) to 100 (best possible), in percent
EQ-Visual Analogue Scale result, at 12 months | 12 months after surgery
  EQ-Visual Analogue Scale, scale 0 (worst) to 100 (best possible), in percent
Results of preoperative Quality of life dimensions | preoperative
  5 dimensions measurable with EQ5D-3L (scale 1,2 or 3) (ordinal scale)
Results of Quality of life dimensions at 6 months after surgery | 6 months after surgery
  5 dimensions measurable with EQ5D-3L (scale 1,2 or 3)(ordinal scale)
Results of Quality of life dimensions at 12 months after surgery | 12 months after surgery
  5 dimensions measurable with EQ5D-3L (scale 1,2 or 3)(ordinal scale)

SECONDARY OUTCOMES:
Overall mortality rate | over the follow-up period ranging 3 to 9 years postoperatively
  Survival after surgery, annual postoperative, in percent
Overall surgical morbidity rate | 0 to 12 months after surgery
  All surgical and cardiovascular complications, in percent

OTHER OUTCOMES:
Re-hospitalization rate | over the follow-up period ranging 3 to 9 years postoperatively
  Re-admittance to health care facilities, annual postoperative, in percent

CONTACTS AND LOCATIONS:
Overall Officials: Jari Laurikka, MD,PhD, Study Director — Head of Department

IPD SHARING:
Plan to Share IPD: No
local legislation prevents personal data sharing